CLINICAL TRIAL: NCT05137236
Title: A Phase 2A, Randomized, Stratified, Observer-Blind Study to Evaluate the Immunogenicity and Safety of mRNA-1283 Vaccine Boosters for SARS-CoV-2
Brief Title: A Study to Evaluate the Immunogenicity and Safety of mRNA-1283 COVID-19 Vaccine Boosters
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1283-P201
Record Dates: First submitted 2021-11-24; First posted 2021-11-30 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A of this study is designed as an observer-blind study. Part B of the study is designed as an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A: mRNA-1283 Dose Level 1 (Experimental): Participants will receive single intramuscular (IM) injection of mRNA-1283 at Dose Level 1 on Day 1.
  Interventions: Biological: mRNA-1283
- Part A: mRNA-1283 Dose Level 2 (Experimental): Participants will receive single IM injection of mRNA-1283 at Dose Level 2 on Day 1.
  Interventions: Biological: mRNA-1283
- Part A: mRNA-1283 Dose Level 3 (Experimental): Participants will receive single IM injection of mRNA-1283 at Dose Level 3 on Day 1.
  Interventions: Biological: mRNA-1283
- Part A: mRNA-1283.211 Dose Level 1 (Experimental): Participants will receive single IM injection of mRNA-1283.211 at Dose Level 1 on Day 1.
  Interventions: Biological: mRNA-1283.211
- Part A: mRNA-1283.211 Dose Level 2 (Experimental): Participants will receive single IM injection of mRNA-1283.211 at Dose Level 2 on Day 1.
  Interventions: Biological: mRNA-1283.211
- Part A: mRNA-1273 (Active Comparator): Participants will receive single IM injection of mRNA-1273 on Day 1.
  Interventions: Biological: mRNA-1273
- Part B: mRNA-1283.529 Dose Level 1 (Experimental): Participants will receive single IM injection of mRNA-1283.529 as a second booster at Dose Level 1 on Day 1.
  Interventions: Biological: mRNA-1283.529
- Part B: mRNA-1283.529 Dose Level 2 (Experimental): Participants will receive single IM injection of mRNA-1283.529 as a second booster at Dose Level 2 on Day 1.
  Interventions: Biological: mRNA-1283.529

INTERVENTIONS:
Biological: mRNA-1283 — Sterile liquid for injection
  Arms: Part A: mRNA-1283 Dose Level 1; Part A: mRNA-1283 Dose Level 2; Part A: mRNA-1283 Dose Level 3
Biological: mRNA-1283.211 — Sterile liquid for injection
  Arms: Part A: mRNA-1283.211 Dose Level 1; Part A: mRNA-1283.211 Dose Level 2
Biological: mRNA-1273 — Sterile liquid for injection
  Arms: Part A: mRNA-1273
Biological: mRNA-1283.529 — Sterile liquid for injection
  Arms: Part B: mRNA-1283.529 Dose Level 1; Part B: mRNA-1283.529 Dose Level 2

SUMMARY:
The main goal of Part A of this study is to assess the safety, reactogenicity, and immunogenicity of the study vaccine candidates. The main goal of Part B of this study is to assess the safety, reactogenicity, and immunogenicity of the mRNA-1283.529 booster vaccine candidate.

DETAILED DESCRIPTION:
Part A of this study will assess whether a single dose of mRNA-1283 at three different dose levels or mRNA-1283.211 at two different dose levels will boost antibody responses to the Wuhan-Hu-1 (ancestral strain of SARS-CoV-2) virus, and to the B.1.351 variant, and potentially other SARS-CoV-2 variants, and it will also be used to select a dose for subsequent clinical evaluation. The study will include an active comparator group of participants who will receive mRNA-1273.

Participants in Part A who received the primary series of mRNA-1273 with appropriate documentation at least 6 months prior will be randomized 1:1:1:1:1:1 to receive a single boost of mRNA-1283 at one of three dose levels, a single boost of mRNA-1283.211 at one of two dose levels, or a single dose of the active comparator, mRNA-1273.

Part B of this study will assess whether a single dose of mRNA-1283.529 at two different dose levels as the second booster after a first booster of mRNA- 1273, at least 3 months prior, will boost antibody response to the ancestral strain of the SARS-CoV-2 virus, the B.1.1.529 variant, and potentially other SARS-CoV-2 variants, and inform dose selection for mRNA-1283.529 booster vaccine candidate for subsequent clinical evaluation.

Participants in Part B who received the primary series of mRNA 1273 and who received a first booster dose of mRNA-1273 at least 3 months prior will be enrolled in a 1:1 ratio to receive a single boost of mRNA 1283.529 at one of two dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of nonchildbearing potential may be enrolled in the study. Nonchildbearing potential is defined as bilateral tubal ligation >1 year prior to screening, bilateral oophorectomy, hysterectomy, or menopause.
* Female participants of childbearing potential may be enrolled in the study if the participant has a negative pregnancy test on the day of vaccination (Day 1), practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, agreed to continue adequate contraception through 3 months following the last vaccine administration, and not currently breastfeeding.
* Participant must have received their second dose of the mRNA-1273 primary series at least 6 months prior to screening and enrollment (Part A) or have received the mRNA-1273 series and an mRNA-1273 booster dose at least 3 months prior to screening and enrollment (Part B).

Exclusion Criteria:

* Had significant exposure to someone with SARS-CoV-2 infection or COVID-19 in the past 14 days, defined by the US Centers for Disease Control and Prevention (CDC) as a close contact of someone who has COVID-19.
* Is acutely ill or febrile (temperature ≥38.0 degree Celsius [°C]/100.4 degree Fahrenheit [°F]) less than 72 hours prior to or at the screening visit or Day 1.
* Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation, or that could interfere with safety assessments or interpretation of results according to the investigator's judgment.
* Has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to screening (for corticosteroids ≥10 milligrams [mg]/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Has received or plans to receive any licensed vaccine ≤28 days prior to the injection (Day 1) or plans to receive a licensed vaccine within 28 days before or after the study injection, with the exception of influenza vaccines, which may be given 14 days before or after receipt of a study vaccine.
* Has received systemic immunoglobulins or blood products within 3 months prior to the screening visit, or plans to receive these during the study.
* Has donated ≥ 450 milliliters (mL) of blood products within 28 days prior to the screening visit or plans to donate blood products during the study.
* Plans to participate in an interventional clinical trial of an investigational vaccine or drug while participating in this study.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - MedPharmics, LLC, Phoenix, Arizona
  - Research Centers of America, Hollywood, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Tekton Research, Chamblee, Georgia
  - MedPharmics, Metairie, Louisiana
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Clinical Research Institute, Inc - CRN, Minneapolis, Minnesota
  - Meridian Clinical Research (Nebraska), Lincoln, Nebraska
  - MedPharmics, LLC. - Albuquerque, Albuquerque, New Mexico
  - Rochester Clinical Research, Inc., Rochester, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Meridian Clinical Research (Cincinnati), Cincinnati, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - ACRC Trials, Frisco, Texas
  - Ventavia Research Group, Houston, Texas
  - Health Research of Hampton Roads Inc., Newport News, Virginia

REFERENCES:
- [Derived] Chalkias S, Pragalos A, Akinsola A, Berman G, Ampajwala M, Meyer J, Schoch L, Zhou W, Paila YD, Deng W, Feng J, de Windt E, Edwards D, Miller J, Das R. Safety and Immunogenicity of SARS-CoV-2 Spike Receptor-Binding Domain and N-Terminal Domain mRNA Vaccine. J Infect Dis. 2025 Apr 15;231(4):e754-e763. doi: 10.1093/infdis/jiaf022. PMID 39792478
- [Derived] Stewart-Jones GBE, Elbashir SM, Wu K, Lee D, Renzi I, Ying B, Koch M, Sein CE, Choi A, Whitener B, Garcia-Dominguez D, Henry C, Woods A, Ma L, Montes Berrueta D, Avena LE, Quinones J, Falcone S, Hsiao CJ, Scheaffer SM, Thackray LB, White P, Diamond MS, Edwards DK, Carfi A. Domain-based mRNA vaccines encoding spike protein N-terminal and receptor binding domains confer protection against SARS-CoV-2. Sci Transl Med. 2023 Sep 13;15(713):eadf4100. doi: 10.1126/scitranslmed.adf4100. Epub 2023 Sep 13. PMID 37703353
- [Derived] Stewart-Jones GBE, Elbashir SM, Wu K, Lee D, Renzi I, Ying B, Koch M, Sein CE, Choi A, Whitener B, Garcia-Dominguez D, Henry C, Woods A, Ma L, Montes Berrueta D, Avena LE, Quinones J, Falcone S, Hsiao CJ, Scheaffer SM, Thackray LB, White P, Diamond MS, Edwards DK, Carfi A. Development of SARS-CoV-2 mRNA vaccines encoding spike N-terminal and receptor binding domains. bioRxiv [Preprint]. 2022 Oct 7:2022.10.07.511319. doi: 10.1101/2022.10.07.511319. PMID 36238717

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow data are reported per initial randomized treatment.
Groups:
- Part A: mRNA-1283 Low Dose: Participants received a single intramuscular (IM) injection of mRNA-1283 at low dose on Day 1.
- Part A: mRNA-1283 Medium Dose: Participants received a single IM injection of mRNA-1283 at medium dose on Day 1.
- Part A: mRNA-1283 High Dose: Participants received a single IM injection of mRNA-1283 at high dose on Day 1.
- Part A: mRNA-1283.211 Low Dose: Participants received a single IM injection of mRNA-1283.211 at low dose on Day 1.
- Part A: mRNA-1283.211 High Dose: Participants received a single IM injection of mRNA-1283.211 at high dose on Day 1.
- Part A: mRNA-1273: Participants received a single IM injection of mRNA-1273 on Day 1.
- Part B: mRNA-1283.529 Low Dose: Participants received a single IM injection of mRNA-1283.529 as a second booster at low dose on Day 1.
- Part B: mRNA-1283.529 High Dose: Participants received a single IM injection of mRNA-1283.529 as a second booster at high dose on Day 1.
Period: Part A
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273 | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Started | 57 | 63 | 56 | 53 | 54 | 57 | 0 (Participants in Part B arms were not enrolled into Part A of the trial.) | 0 (Participants in Part B arms were not enrolled into Part A of the trial.)
Received at Least 1 Dose of Study Drug | 57 | 63 | 56 | 53 (One participant in the mRNA-1283.211 low dose group had a dosing error and received mRNA-1283 at medium dose.) | 54 | 57 | 0 | 0
Completed | 51 | 52 | 54 | 49 | 48 | 47 | 0 | 0
Not Completed | 6 | 11 | 2 | 4 | 6 | 10 | 0 | 0
Not completed — Other than Specified | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 1 | 1 | 3 | 2 | 0 | 0
Not completed — Lost to Follow-up | 5 | 7 | 1 | 3 | 3 | 8 | 0 | 0
Period: Part B
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273 | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Started | 0 (Participants in Part A arms were not enrolled into Part B of the trial.) | 0 (Participants in Part A arms were not enrolled into Part B of the trial.) | 0 (Participants in Part A arms were not enrolled into Part B of the trial.) | 0 (Participants in Part A arms were not enrolled into Part B of the trial.) | 0 (Participants in Part A arms were not enrolled into Part B of the trial.) | 0 (Participants in Part A arms were not enrolled into Part B of the trial.) | 103 | 97
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 103 | 97
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 98 | 88
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Measured in the Safety Set, which consisted of all randomized/enrolled (Part A: randomized, Part B: enrolled) participants who received one dose of investigational product (IP). Data in the Safety Set is presented per actual dose received. There was 1 participant in the mRNA-1283.211 low dose group who had a dosing error and received mRNA-1283 at medium dose.
Groups:
- Part A: mRNA-1283 Low Dose: Participants received a single IM injection of mRNA-1283 at low dose on Day 1.
- Total: Total of all reporting groups
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273 | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose | Total
Number analyzed (Participants) | 57 | 64 | 56 | 52 | 54 | 57 | 103 | 97 | 540
Age, Customized [Count of Participants; unit: Participants]
  >=18 and <56 Years | 40 | 46 | 42 | 37 | 40 | 42 | 44 | 59 | 350
  >=56 Years | 17 | 18 | 14 | 15 | 14 | 15 | 59 | 38 | 190
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 43 | 32 | 34 | 39 | 32 | 70 | 62 | 343
  Male | 26 | 21 | 24 | 18 | 15 | 25 | 33 | 35 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 14 | 8 | 9 | 8 | 11 | 2 | 4 | 66
  Not Hispanic or Latino | 47 | 50 | 47 | 43 | 43 | 45 | 100 | 93 | 468
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3
  Asian | 5 | 1 | 3 | 3 | 3 | 3 | 0 | 2 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 11 | 11 | 9 | 9 | 10 | 6 | 7 | 7 | 70
  White | 41 | 48 | 41 | 38 | 37 | 47 | 94 | 88 | 434
  More than one race | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 6
  Unknown or Not Reported | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Parts A and B: Number of Participants With Solicited Local and Solicited Systemic Reactogenicity Adverse Reactions (ARs)
Description: An AR is any adverse event (AE) related to the IP injection. Solicited local ARs included pain at injection site, erythema (redness) at injection site, swelling (hardness) at injection site, localized axillary swelling or tenderness ipsilateral to the injection arm, and groin or underarm swelling or tenderness ipsilateral to the side of injection. Solicited systemic ARs included headache, fatigue, myalgia (muscle aches all over the body), arthralgia (aching in several joints), nausea/vomiting, fever, chills, irritability/crying, sleepiness, and loss of appetite. Note, not all solicited ARs were considered AEs. The Investigator determined if solicited AR was also to be recorded as an AE. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to Day 7
Population: Measured in the Solicited Safety Set, which consisted of all participants in the Safety Set who contributed any solicited AR data.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273 | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 54 | 60 | 52 | 48 | 46 | 54 | 103 | 96
Participants
  Solicited Local ARs | 30 | 40 | 37 | 28 | 29 | 46 | 46 | 69
  Solicited Systemic ARs | 32 | 39 | 35 | 39 | 27 | 41 | 51 | 60

2. Primary Outcome: Parts A and B: Number of Participants With Unsolicited AEs
Description: An unsolicited AE was defined as any AE reported by the participant that was not specified as a solicited AR in the protocol or was specified as a solicited AR but started outside the protocol-defined period for reporting solicited ARs. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to Day 28
Population: Measured in the Safety Set, which consisted of all randomized/enrolled (Part A: randomized, Part B: enrolled) participants who received one dose of IP. Data in the Safety Set is presented per actual dose received. There was 1 participant in the mRNA-1283.211 low dose group who had a dosing error and received mRNA-1283 at medium dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273 | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 57 | 64 | 56 | 52 | 54 | 57 | 103 | 97
Participants | 13 | 9 | 11 | 12 | 7 | 8 | 13 | 11

3. Primary Outcome: Parts A and B: Number of Participants With Serious Adverse Events (SAEs), Medically Attended AEs (MAAEs), AEs Leading to Withdrawal From Study Participation and AEs of Special Interest (AESIs)
Description: SAEs were AEs that resulted in death, were life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, a congenital anomaly or birth defect, or was a medically important event. MAAEs were AEs that lead to an unscheduled visit to a healthcare provider. AESIs were AEs (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program for which ongoing monitoring and immediate notification by the investigator to the Sponsor was required. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Day 1 to Day 366
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273 | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 57 | 64 | 56 | 52 | 54 | 57 | 103 | 97
Participants
  SAEs | 2 | 1 | 2 | 3 | 3 | 2 | 2 | 6
  MAAEs | 25 | 23 | 27 | 24 | 18 | 23 | 51 | 42
  AEs Leading to Withdrawal from Study Participation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  AESIs | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3

4. Primary Outcome: Part A: Geometric Mean Titer (GMT) of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Specific Neutralizing Antibody (nAb) Against Ancestral SARS-CoV-2 and Against SARS-CoV-2 Variant B.1.351
Description: The GMT (50% inhibitory dose [ID50]) of nAb against ancestral SARS-CoV-2 and against SARS-CoV-2 variant B.1.351 are reported.
Time Frame: Day 29
Population: Measured in the Per-Protocol Set for Immunogenicity - Pre-booster SARS-CoV-2 Negative, which consisted of all participants in the full analysis set (FAS) who received the planned dose of IP and who had no major protocol deviations that impact key or critical data who were pre-booster SARS-CoV-2 negative and had evaluable data for the endpoint. Here, number analyzed signifies those participants who were evaluable for specified categories only.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273
Number analyzed (Participants) | 31 | 38 | 32 | 24 | 22 | 28
Titer
  Ancestral SARS-CoV-2 ID50 | 4751.7 [3207.0 to 7040.5] | 5666.5 [4149.3 to 7738.4] | 7723.0 [5621.7 to 10609.7] | 5105.5 [3083.3 to 8453.9] | 4729.8 [2572.4 to 8696.3] | 3562.9 [2550.1 to 4977.9]
  SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 38 | 32 | 24 | 22 | 28
  SARS-CoV-2 Variant B.1.351 ID50 | 946.7 [611.4 to 1465.7] | 1216.2 [838.9 to 1763.3] | 2020.1 [1350.7 to 3021.1] | 1566.3 [942.4 to 2603.2] | 1224.8 [660.6 to 2271.0] | 964.4 [659.6 to 1410.1]

5. Primary Outcome: Part A: Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Specific nAb Against Ancestral SARS-CoV-2 and Against SARS-CoV-2 Variant B.1.351
Description: The GMFR measures the changes in immunogenicity titers or levels within participants.
Time Frame: Day 29
Population: Measured in the Per-Protocol Set for Immunogenicity - Pre-booster SARS-CoV-2 Negative, which consisted of all participants in the FAS who received the planned dose of IP and who had no major protocol deviations that impact key or critical data who were pre-booster SARS-CoV-2 negative and had evaluable data for the endpoint. Here, number analyzed signifies those participants who were evaluable for specified categories only.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273
Number analyzed (Participants) | 31 | 38 | 32 | 24 | 22 | 28
Ratio
  Ancestral SARS-CoV-2 ID50 | 26.8 [16.8 to 42.8] | 34.3 [20.9 to 56.0] | 45.3 [27.0 to 76.0] | 35.5 [18.1 to 69.6] | 28.1 [13.2 to 59.9] | 24.5 [14.7 to 40.7]
  SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 38 | 32 | 24 | 22 | 28
  SARS-CoV-2 Variant B.1.351 ID50 | 27.4 [16.2 to 46.6] | 33.7 [21.1 to 53.9] | 52.1 [30.2 to 89.8] | 54.2 [27.2 to 107.7] | 41.8 [20.8 to 84.0] | 35.8 [19.8 to 64.6]

6. Primary Outcome: Part A: Number of Participants With Seroresponse Against Ancestral SARS-CoV-2 and Against SARS-CoV-2 Variant B.1.351
Description: Seroresponse was defined as an increase of SARS-CoV-2 specific binding antibody (bAb) level or nAb titer to at least 4x lower limit of quantification (LLOQ) if the baseline is below the LLOQ, or a 4-fold or greater rise if pre-booster ≥ LLOQ.
Time Frame: Day 29
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273
Number analyzed (Participants) | 31 | 38 | 32 | 24 | 22 | 28
Participants
  Ancestral SARS-CoV-2 ID50 | 28 | 35 | 30 | 22 | 19 | 26
  SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 38 | 32 | 24 | 22 | 28
  SARS-CoV-2 Variant B.1.351 ID50 | 26 | 35 | 31 | 22 | 19 | 25

7. Primary Outcome: Part B: GMT of SARS-CoV-2 Specific nAb Against SARS-CoV-2 Omicron Variant (B.1.1.529)
Description: The GMT (ID50) of nAb against SARS-CoV-2 omicron variant (B.1.1.529) are reported.
Time Frame: Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 75 | 69
Titer | 1562.9 [1113.4 to 2194.0] | 2723.0 [1938.3 to 3825.4]

8. Primary Outcome: Part B: GMFR of SARS-CoV-2 Specific nAb Against SARS-CoV-2 Omicron Variant (B.1.1.529)
Description: The GMFR measures the changes in immunogenicity titers or levels within participants.
Time Frame: Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 75 | 69
Ratio | 7.2 [5.7 to 9.0] | 7.8 [5.9 to 10.4]

9. Primary Outcome: Part B: Number of Participants With Seroresponse Against SARS-CoV-2 Omicron Variant (B.1.1.529)
Description: Seroresponse was defined as an increase of SARS-CoV-2 specific bAb level or nAb titer to at least 4x LLOQ if the baseline is below the LLOQ, or a 4-fold or greater rise if pre-booster ≥ LLOQ.
Time Frame: Day 29
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 75 | 69
Participants | 55 | 48

10. Secondary Outcome: Part A: GMT of SARS-CoV-2 Specific nAb Against Ancestral SARS-CoV-2 and Against SARS-CoV-2 Variant B.1.351
Description: The GMT (ID50) of nAb against ancestral SARS-CoV-2 and against SARS-CoV-2 Variant B.1.351 are reported.
Time Frame: Days 1, 29, 91, 181, and 366
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273
Number analyzed (Participants) | 31 | 38 | 32 | 24 | 22 | 28
Titer
  Day 1 Ancestral SARS-CoV-2 ID50 | 177.4 [108.5 to 290.0] | 165.4 [114.4 to 239.2] | 170.4 [104.4 to 278.0] | 143.7 [97.0 to 213.1] | 168.6 [74.5 to 381.3] | 145.6 [91.9 to 230.7]
  Day 29 Ancestral SARS-CoV-2 ID50 | 4751.7 [3207.0 to 7040.5] | 5666.5 [4149.3 to 7738.4] | 7723.0 [5621.7 to 10609.7] | 5105.5 [3083.3 to 8453.9] | 4729.8 [2572.4 to 8696.3] | 3562.9 [2550.1 to 4977.9]
  Day 91 Ancestral SARS-CoV-2 ID50: number analyzed (Participants) | 31 | 36 | 32 | 23 | 22 | 28
  Day 91 Ancestral SARS-CoV-2 ID50 | 3980.4 [2459.2 to 6442.6] | 4589.2 [3285.9 to 6409.4] | 6754.5 [4604.3 to 9909.0] | 4943.1 [3029.0 to 8066.9] | 4319.8 [2758.9 to 6763.7] | 3155.1 [1980.2 to 5027.0]
  Day 181 Ancestral SARS-CoV-2 ID50: number analyzed (Participants) | 30 | 36 | 31 | 24 | 21 | 26
  Day 181 Ancestral SARS-CoV-2 ID50 | 2476.4 [1400.5 to 4378.8] | 2861.4 [1879.2 to 4357.1] | 3834.7 [2606.2 to 5642.2] | 2960.3 [1805.5 to 4853.6] | 2767.2 [1588.2 to 4821.6] | 1269.4 [809.8 to 1990.0]
  Day 366 Ancestral SARS-CoV-2 ID50: number analyzed (Participants) | 26 | 29 | 30 | 21 | 19 | 22
  Day 366 Ancestral SARS-CoV-2 ID50 | 1497.4 [723.2 to 3100.5] | 3097.6 [2003.1 to 4790.2] | 2921.1 [2062.2 to 4137.8] | 2013.3 [1225.1 to 3308.5] | 1539.6 [772.8 to 3067.3] | 1336.1 [739.4 to 2414.2]
  Day 1 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 38 | 32 | 24 | 22 | 27
  Day 1 SARS-CoV-2 Variant B.1.351 ID50 | 34.5 [21.0 to 56.5] | 36.1 [25.9 to 50.3] | 38.8 [24.0 to 62.6] | 28.9 [19.0 to 44.0] | 29.3 [14.2 to 60.4] | 27.9 [17.5 to 44.6]
  Day 29 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 38 | 32 | 24 | 22 | 28
  Day 29 SARS-CoV-2 Variant B.1.351 ID50 | 946.7 [611.4 to 1465.7] | 1216.2 [838.9 to 1763.3] | 2020.1 [1350.7 to 3021.1] | 1566.3 [942.4 to 2603.2] | 1224.8 [660.6 to 2271.0] | 964.4 [659.6 to 1410.1]
  Day 91 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 36 | 32 | 23 | 22 | 28
  Day 91 SARS-CoV-2 Variant B.1.351 ID50 | 794.8 [461.9 to 1367.5] | 965.6 [631.0 to 1477.7] | 1520.8 [1025.7 to 2254.8] | 1105.8 [579.9 to 2108.6] | 990.5 [591.0 to 1660.0] | 640.2 [384.2 to 1066.7]
  Day 181 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 36 | 31 | 24 | 21 | 26
  Day 181 SARS-CoV-2 Variant B.1.351 ID50 | 786.3 [403.1 to 1533.7] | 760.2 [438.7 to 1317.2] | 1458.4 [916.6 to 2320.5] | 967.2 [531.3 to 1760.7] | 769.6 [429.6 to 1378.9] | 460.5 [266.1 to 796.9]
  Day 366 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 25 | 29 | 30 | 21 | 19 | 22
  Day 366 SARS-CoV-2 Variant B.1.351 ID50 | 581.2 [279.7 to 1207.6] | 1461.8 [855.0 to 2499.1] | 1259.6 [789.7 to 2009.1] | 790.3 [397.0 to 1573.3] | 530.3 [223.4 to 1258.4] | 534.2 [252.1 to 1132.1]

11. Secondary Outcome: Part A: GMT of SARS-CoV-2 Specific bAb Against Ancestral SARS-CoV-2 and Against SARS-CoV-2 Variant B.1.351
Description: The GMT of bAb against ancestral SARS-CoV-2 and against SARS-CoV-2 Variant B.1.351 are reported.
Time Frame: Days 1, 29, 91, 181, and 366
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273
Number analyzed (Participants) | 31 | 38 | 32 | 24 | 22 | 28
Titer
  Day 1 Ancestral SARS-CoV-2: number analyzed (Participants) | 30 | 38 | 32 | 24 | 22 | 27
  Day 1 Ancestral SARS-CoV-2 | 29458.4 [18988.8 to 45700.5] | 29839.6 [21775.9 to 40889.2] | 32632.4 [22347.8 to 47650.0] | 28886.5 [21389.0 to 39012.1] | 30803.7 [17375.8 to 54608.8] | 30644.3 [21431.7 to 43817.0]
  Day 29 Ancestral SARS-CoV-2: number analyzed (Participants) | 30 | 38 | 32 | 24 | 22 | 28
  Day 29 Ancestral SARS-CoV-2 | 717040.9 [545647.9 to 942269.9] | 737925.6 [580477.3 to 938080.1] | 1070144.5 [823120.1 to 1391302.9] | 835783.7 [570117.5 to 1225246.2] | 688909.2 [429957.5 to 1103820.5] | 594926.9 [462362.9 to 765498.3]
  Day 91 Ancestral SARS-CoV-2: number analyzed (Participants) | 31 | 36 | 32 | 23 | 22 | 28
  Day 91 Ancestral SARS-CoV-2 | 538518.6 [370446.8 to 782844.8] | 575062.5 [432778.8 to 764124.4] | 785822.0 [601645.3 to 1026379.3] | 613915.9 [398665.6 to 945385.7] | 629867.6 [446549.5 to 888441.8] | 390985.5 [289339.3 to 528340.5]
  Day 181 Ancestral SARS-CoV-2: number analyzed (Participants) | 30 | 35 | 30 | 24 | 20 | 26
  Day 181 Ancestral SARS-CoV-2 | 349027.0 [227163.4 to 536265.3] | 338163.9 [239965.4 to 476547.2] | 447634.3 [336503.1 to 595467.0] | 370694.6 [257195.7 to 534280.0] | 358399.9 [238972.0 to 537512.6] | 198042.8 [141579.1 to 277025.1]
  Day 366 Ancestral SARS-CoV-2: number analyzed (Participants) | 26 | 29 | 30 | 21 | 19 | 22
  Day 366 Ancestral SARS-CoV-2 | 220315.4 [125437.1 to 386957.9] | 390137.4 [266323.9 to 571511.7] | 370475.8 [277402.5 to 494776.9] | 260942.1 [185711.7 to 366647.8] | 246749.8 [150746.4 to 403893.4] | 163960.1 [107650.0 to 249725.1]
  Day 1 SARS-CoV-2 Variant B.1.351: number analyzed (Participants) | 25 | 33 | 25 | 17 | 17 | 23
  Day 1 SARS-CoV-2 Variant B.1.351 | 12499.8 [8275.5 to 18880.3] | 13289.6 [9765.0 to 18086.4] | 15875.3 [10891.6 to 23139.3] | 15255.0 [10255.8 to 22691.2] | 12664.6 [7792.9 to 20581.8] | 17401.8 [11236.5 to 26950.0]
  Day 29 SARS-CoV-2 Variant B.1.351: number analyzed (Participants) | 25 | 33 | 25 | 17 | 17 | 24
  Day 29 SARS-CoV-2 Variant B.1.351 | 359208.1 [259502.7 to 497221.9] | 369055.6 [277237.5 to 491282.7] | 504673.7 [387088.6 to 657977.5] | 399270.2 [261474.1 to 609684.5] | 352867.0 [193718.3 to 642763.9] | 333866.2 [264529.3 to 421377.3]
  Day 91 SARS-CoV-2 Variant B.1.351: number analyzed (Participants) | 26 | 31 | 25 | 16 | 17 | 24
  Day 91 SARS-CoV-2 Variant B.1.351 | 237940.9 [154308.2 to 366901.3] | 271701.9 [194943.5 to 378683.7] | 362689.3 [275141.6 to 478093.9] | 245501.5 [154897.5 to 389102.6] | 330103.6 [246861.3 to 441415.5] | 202152.0 [158047.0 to 258564.9]
  Day 181 SARS-CoV-2 Variant B.1.351: number analyzed (Participants) | 26 | 30 | 23 | 17 | 15 | 22
  Day 181 SARS-CoV-2 Variant B.1.351 | 151202.9 [90854.0 to 251638.2] | 143620.7 [94068.8 to 219274.8] | 184376.3 [134452.0 to 252838.3] | 142996.2 [92494.0 to 221072.9] | 183952.8 [130226.4 to 259844.8] | 95496.2 [70938.4 to 128555.5]
  Day 366 SARS-CoV-2 Variant B.1.351: number analyzed (Participants) | 23 | 25 | 23 | 14 | 14 | 19
  Day 366 SARS-CoV-2 Variant B.1.351 | 105204.5 [53545.8 to 206701.3] | 218574.3 [128094.7 to 372964.0] | 203600.7 [133854.9 to 309687.7] | 121911.8 [68950.3 to 215553.6] | 134120.4 [70688.7 to 254471.9] | 89012.3 [53840.6 to 147160.1]

12. Secondary Outcome: Part B: GMT of SARS-CoV-2 Specific nAb Against SARS-CoV-2 Omicron Variant (B.1.1.529)
Description: The GMT (ID50) of nAb against SARS-CoV-2 omicron variant (B.1.1.529) are reported.
Time Frame: Days 1, 29, 91, 181, and 366
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 75 | 69
Titer
  Day 1 SARS-CoV-2 Variant B.1.1.529 ID50 | 217.6 [162.0 to 292.4] | 349.2 [239.7 to 508.7]
  Day 29 SARS-CoV-2 Variant B.1.1.529 ID50 | 1562.9 [1113.4 to 2194.0] | 2723.0 [1938.3 to 3825.4]
  Day 91 SARS-CoV-2 Variant B.1.1.529 ID50: number analyzed (Participants) | 73 | 66
  Day 91 SARS-CoV-2 Variant B.1.1.529 ID50 | 978.5 [667.7 to 1434.0] | 1713.5 [1238.2 to 2371.4]
  Day 181 SARS-CoV-2 Variant B.1.1.529 ID50: number analyzed (Participants) | 73 | 64
  Day 181 SARS-CoV-2 Variant B.1.1.529 ID50 | 724.0 [500.9 to 1046.5] | 1608.7 [1053.9 to 2455.5]
  Day 366 SARS-CoV-2 Variant B.1.1.529 ID50: number analyzed (Participants) | 43 | 39
  Day 366 SARS-CoV-2 Variant B.1.1.529 ID50 | 666.0 [395.5 to 1121.8] | 1873.7 [1156.9 to 3034.9]

13. Secondary Outcome: Part B: GMT of SARS-CoV-2 Specific bAb Against SARS-CoV-2 Omicron Variant (B.1.1.529)
Description: The GMT of bAb against SARS-CoV-2 omicron variant (B.1.1.529) are reported.
Time Frame: Days 1, 29, 91, 181, and 366
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 74 | 67
Titer
  Day 1 SARS-CoV-2 Variant B.1.1.529 | 50830.3 [41890.8 to 61677.5] | 61419.3 [49407.6 to 76351.2]
  Day 29 SARS-CoV-2 Variant B.1.1.529 | 182046.9 [153016.2 to 216585.4] | 233677.5 [189382.6 to 288332.8]
  Day 91 SARS-CoV-2 Variant B.1.1.529: number analyzed (Participants) | 72 | 61
  Day 91 SARS-CoV-2 Variant B.1.1.529 | 118658.1 [97721.5 to 144080.3] | 157262.3 [126717.0 to 195170.7]
  Day 181 SARS-CoV-2 Variant B.1.1.529: number analyzed (Participants) | 72 | 63
  Day 181 SARS-CoV-2 Variant B.1.1.529 | 73469.5 [58947.0 to 91569.8] | 103322.9 [81221.9 to 131437.7]
  Day 366 SARS-CoV-2 Variant B.1.1.529: number analyzed (Participants) | 42 | 39
  Day 366 SARS-CoV-2 Variant B.1.1.529 | 46721.5 [32757.5 to 66638.1] | 98989.7 [67965.4 to 144175.8]

14. Secondary Outcome: Part A: GMFR of SARS-CoV-2 Specific nAb Against Ancestral SARS-CoV-2 and Against SARS-CoV-2 Variant B.1.351
Description: The GMFR measures the changes in immunogenicity titers or levels within participants.
Time Frame: Days 29, 91, 181, and 366
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273
Number analyzed (Participants) | 31 | 38 | 32 | 24 | 22 | 28
Ratio
  Day 29 Ancestral SARS-CoV-2 ID50 | 26.8 [16.8 to 42.8] | 34.3 [20.9 to 56.0] | 45.3 [27.0 to 76.0] | 35.5 [18.1 to 69.6] | 28.1 [13.2 to 59.9] | 24.5 [14.7 to 40.7]
  Day 91 Ancestral SARS-CoV-2 ID50: number analyzed (Participants) | 31 | 36 | 32 | 23 | 22 | 28
  Day 91 Ancestral SARS-CoV-2 ID50 | 22.4 [13.5 to 37.4] | 27.1 [16.5 to 44.6] | 39.6 [23.0 to 68.3] | 34.0 [17.2 to 67.1] | 25.6 [12.2 to 53.9] | 21.7 [12.4 to 38.0]
  Day 181 Ancestral SARS-CoV-2 ID50: number analyzed (Participants) | 30 | 36 | 31 | 24 | 21 | 26
  Day 181 Ancestral SARS-CoV-2 ID50 | 13.9 [7.4 to 26.0] | 17.1 [9.9 to 29.7] | 23.6 [13.2 to 42.1] | 20.6 [11.1 to 38.2] | 15.3 [7.6 to 30.7] | 8.2 [4.6 to 14.6]
  Day 366 Ancestral SARS-CoV-2 ID50: number analyzed (Participants) | 26 | 29 | 30 | 21 | 19 | 22
  Day 366 Ancestral SARS-CoV-2 ID50 | 9.1 [4.3 to 19.2] | 18.0 [9.5 to 33.9] | 17.8 [10.3 to 30.6] | 13.7 [7.1 to 26.4] | 9.8 [4.1 to 23.3] | 8.7 [4.3 to 17.6]
  Day 29 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 38 | 32 | 24 | 22 | 27
  Day 29 SARS-CoV-2 Variant B.1.351 ID50 | 27.4 [16.2 to 46.6] | 33.7 [21.1 to 53.9] | 52.1 [30.2 to 89.8] | 54.2 [27.2 to 107.7] | 41.8 [20.8 to 84.0] | 35.8 [19.8 to 64.6]
  Day 91 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 36 | 32 | 23 | 22 | 27
  Day 91 SARS-CoV-2 Variant B.1.351 ID50 | 23.0 [12.8 to 41.6] | 27.0 [16.5 to 44.4] | 39.2 [21.9 to 70.3] | 38.1 [16.9 to 85.9] | 33.8 [17.7 to 64.6] | 23.9 [12.7 to 45.3]
  Day 181 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 29 | 36 | 31 | 24 | 21 | 25
  Day 181 SARS-CoV-2 Variant B.1.351 ID50 | 21.4 [10.1 to 45.1] | 21.4 [12.3 to 37.2] | 39.3 [21.0 to 73.4] | 33.4 [15.8 to 70.6] | 24.9 [12.6 to 49.4] | 16.5 [8.3 to 32.8]
  Day 366 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 24 | 29 | 30 | 21 | 19 | 21
  Day 366 SARS-CoV-2 Variant B.1.351 ID50 | 17.6 [8.0 to 38.7] | 38.2 [20.0 to 73.2] | 32.5 [17.6 to 59.7] | 27.4 [12.3 to 61.0] | 20.0 [7.9 to 50.4] | 18.9 [8.0 to 44.7]

15. Secondary Outcome: Part A: GMFR of SARS-CoV-2 Specific bAb Against Ancestral SARS-CoV-2 and Against SARS-CoV-2 Variant B.1.351
Description: The GMFR measures the changes in immunogenicity titers or levels within participants.
Time Frame: Days 29, 91, 181, and 366
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273
Number analyzed (Participants) | 31 | 38 | 32 | 24 | 22 | 28
Ratio
  Day 29 Ancestral SARS-CoV-2: number analyzed (Participants) | 30 | 38 | 32 | 24 | 22 | 27
  Day 29 Ancestral SARS-CoV-2 | 24.3 [16.1 to 36.9] | 24.7 [16.2 to 37.7] | 32.8 [21.4 to 50.2] | 28.9 [16.2 to 51.6] | 22.4 [12.1 to 41.4] | 19.8 [12.4 to 31.4]
  Day 91 Ancestral SARS-CoV-2: number analyzed (Participants) | 30 | 36 | 32 | 23 | 22 | 27
  Day 91 Ancestral SARS-CoV-2 | 17.5 [11.3 to 27.2] | 19.0 [12.1 to 29.8] | 24.1 [15.6 to 37.3] | 20.9 [11.3 to 38.5] | 20.4 [12.2 to 34.3] | 12.8 [8.2 to 20.0]
  Day 181 Ancestral SARS-CoV-2: number analyzed (Participants) | 29 | 35 | 30 | 24 | 20 | 25
  Day 181 Ancestral SARS-CoV-2 | 11.5 [7.1 to 18.7] | 11.2 [6.9 to 18.2] | 14.0 [8.8 to 22.3] | 12.8 [7.6 to 21.8] | 11.6 [6.8 to 20.0] | 6.2 [3.9 to 9.9]
  Day 366 Ancestral SARS-CoV-2: number analyzed (Participants) | 25 | 29 | 30 | 21 | 19 | 21
  Day 366 Ancestral SARS-CoV-2 | 8.5 [4.8 to 15.0] | 12.9 [7.5 to 22.1] | 11.4 [7.4 to 17.5] | 8.8 [5.3 to 14.8] | 8.5 [4.5 to 16.1] | 5.3 [3.0 to 9.4]
  Day 29 SARS-CoV-2 Variant B.1.351: number analyzed (Participants) | 25 | 33 | 25 | 17 | 17 | 23
  Day 29 SARS-CoV-2 Variant B.1.351 | 28.7 [18.9 to 43.8] | 27.8 [17.6 to 43.8] | 31.8 [20.3 to 49.8] | 26.2 [14.1 to 48.7] | 27.9 [13.1 to 59.4] | 19.8 [12.0 to 32.7]
  Day 91 SARS-CoV-2 Variant B.1.351: number analyzed (Participants) | 25 | 31 | 25 | 16 | 17 | 23
  Day 91 SARS-CoV-2 Variant B.1.351 | 18.1 [11.4 to 28.7] | 20.5 [12.7 to 33.1] | 22.8 [14.0 to 37.4] | 15.9 [8.1 to 31.0] | 26.1 [15.1 to 45.0] | 11.7 [7.5 to 18.3]
  Day 181 SARS-CoV-2 Variant B.1.351: number analyzed (Participants) | 25 | 30 | 23 | 17 | 15 | 21
  Day 181 SARS-CoV-2 Variant B.1.351 | 11.5 [6.8 to 19.6] | 10.8 [6.3 to 18.4] | 11.9 [7.1 to 20.0] | 9.4 [5.2 to 17.0] | 15.0 [8.5 to 26.6] | 5.1 [3.2 to 8.2]
  Day 366 SARS-CoV-2 Variant B.1.351: number analyzed (Participants) | 22 | 25 | 23 | 14 | 14 | 18
  Day 366 SARS-CoV-2 Variant B.1.351 | 8.3 [4.4 to 16.0] | 17.1 [9.4 to 31.1] | 12.9 [7.6 to 21.7] | 7.7 [3.4 to 17.5] | 12.4 [6.0 to 25.5] | 5.2 [2.7 to 9.8]

16. Secondary Outcome: Part B: GMFR of SARS-CoV-2 Specific nAb Against SARS-CoV-2 Omicron Variant (B.1.1.529)
Description: The GMFR measures the changes in immunogenicity titers or levels within participants.
Time Frame: Days 29, 91, 181, and 366
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 75 | 69
Ratio
  Day 29 SARS-CoV-2 Variant B.1.1.529 ID50 | 7.2 [5.7 to 9.0] | 7.8 [5.9 to 10.4]
  Day 91 SARS-CoV-2 Variant B.1.1.529 ID50: number analyzed (Participants) | 73 | 66
  Day 91 SARS-CoV-2 Variant B.1.1.529 ID50 | 4.6 [3.3 to 6.3] | 5.0 [3.6 to 6.8]
  Day 181 SARS-CoV-2 Variant B.1.1.529 ID50: number analyzed (Participants) | 73 | 64
  Day 181 SARS-CoV-2 Variant B.1.1.529 ID50 | 3.4 [2.3 to 5.0] | 4.5 [2.8 to 7.3]
  Day 366 SARS-CoV-2 Variant B.1.1.529 ID50: number analyzed (Participants) | 43 | 39
  Day 366 SARS-CoV-2 Variant B.1.1.529 ID50 | 2.5 [1.5 to 4.3] | 6.4 [3.3 to 12.6]

17. Secondary Outcome: Part B: GMFR of SARS-CoV-2 Specific bAb Against SARS-CoV-2 Omicron Variant (B.1.1.529)
Description: The GMFR measures the changes in immunogenicity titers or levels within participants.
Time Frame: Days 29, 91, 181, and 366
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 74 | 67
Ratio
  Day 29 | 3.6 [3.0 to 4.3] | 3.8 [3.2 to 4.5]
  Day 91: number analyzed (Participants) | 72 | 61
  Day 91 | 2.3 [1.9 to 2.8] | 2.5 [2.0 to 3.0]
  Day 181: number analyzed (Participants) | 72 | 63
  Day 181 | 1.5 [1.2 to 1.8] | 1.6 [1.3 to 2.0]
  Day 366: number analyzed (Participants) | 42 | 39
  Day 366 | 0.9 [0.6 to 1.2] | 1.7 [1.1 to 2.6]

18. Secondary Outcome: Part A: Number of Participants With Seroresponse Against Ancestral SARS-CoV-2 and Against SARS-CoV-2 Variant B.1.351
Description: as for outcome 9
Time Frame: Days 29, 91, 181, and 366
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273
Number analyzed (Participants) | 31 | 38 | 32 | 24 | 22 | 28
Participants
  Day 29 Ancestral SARS-CoV-2 ID50 | 28 | 35 | 30 | 22 | 19 | 26
  Day 91 Ancestral SARS-CoV-2 ID50: number analyzed (Participants) | 31 | 36 | 32 | 23 | 22 | 28
  Day 91 Ancestral SARS-CoV-2 ID50 | 27 | 32 | 29 | 20 | 19 | 26
  Day 181 Ancestral SARS-CoV-2 ID50: number analyzed (Participants) | 30 | 36 | 31 | 24 | 21 | 26
  Day 181 Ancestral SARS-CoV-2 ID50 | 24 | 29 | 27 | 19 | 17 | 17
  Day 366 Ancestral SARS-CoV-2 ID50: number analyzed (Participants) | 26 | 29 | 30 | 21 | 19 | 22
  Day 366 Ancestral SARS-CoV-2 ID50 | 18 | 25 | 27 | 18 | 12 | 14
  Day 29 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 38 | 32 | 24 | 22 | 28
  Day 29 SARS-CoV-2 Variant B.1.351 ID50 | 26 | 35 | 31 | 22 | 19 | 25
  Day 91 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 36 | 32 | 23 | 22 | 28
  Day 91 SARS-CoV-2 Variant B.1.351 ID50 | 26 | 33 | 29 | 20 | 20 | 24
  Day 181 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 30 | 36 | 31 | 24 | 21 | 26
  Day 181 SARS-CoV-2 Variant B.1.351 ID50 | 23 | 30 | 28 | 22 | 17 | 20
  Day 366 SARS-CoV-2 Variant B.1.351 ID50: number analyzed (Participants) | 25 | 29 | 30 | 21 | 19 | 22
  Day 366 SARS-CoV-2 Variant B.1.351 ID50 | 17 | 27 | 28 | 17 | 14 | 16

19. Secondary Outcome: Part B: Number of Participants With Seroresponse Against SARS-CoV-2 Omicron Variant (B.1.1.529)
Description: as for outcome 9
Time Frame: Days 29, 91, 181, and 366
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 75 | 69
Participants
  Day 29 ID50 | 55 | 48
  Day 91 ID50: number analyzed (Participants) | 73 | 66
  Day 91 ID50 | 32 | 35
  Day 181 ID50: number analyzed (Participants) | 73 | 64
  Day 181 ID50 | 26 | 28
  Day 366 ID50: number analyzed (Participants) | 43 | 39
  Day 366 ID50 | 20 | 24

20. Other Pre Specified Outcome: Number of Deaths Related to Study Drug
Description: A death that occurred during the study or that came to the attention of the investigator during the study was reported to the Sponsor, whether or not it was considered related to study drug. The investigator assessed causality (that is, whether there is a reasonable possibility that the study drug caused the death). The relationship was characterized using the following classifications: Not related: There was not a reasonable possibility of a relationship to the study drug. The temporal sequence of the death relative to administration of the study drug was not reasonable AND/OR the death was more likely explained by a cause other than the study drug. Related: There was a reasonable possibility of a relationship to the study drug. There was evidence of exposure to the study drug. The temporal sequence of the death relative to the administration of the study drug was reasonable. The death was more likely explained by the study drug than by another cause.
Time Frame: Day 1 to Day 366
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: mRNA-1283 Low Dose | Part A: mRNA-1283 Medium Dose | Part A: mRNA-1283 High Dose | Part A: mRNA-1283.211 Low Dose | Part A: mRNA-1283.211 High Dose | Part A: mRNA-1273 | Part B: mRNA-1283.529 Low Dose | Part B: mRNA-1283.529 High Dose
Number analyzed (Participants) | 57 | 64 | 56 | 52 | 54 | 57 | 103 | 97
Participants
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Deaths related to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 366
Description: Measured in the Safety Set, which consisted of all randomized/enrolled (Part A: randomized, Part B: enrolled) participants who received one dose of IP. Data in the Safety Set is presented per actual dose received. There was 1 participant in the mRNA-1283.211 low dose group who had a dosing error and received mRNA-1283 at medium dose.
Groups:
- Part A: mRNA-1283 2.5ug Booster: Participants received a single booster dose of mRNA-1283 2.5 ug by intramuscular (IM) injection on day 1
- Part A: mRNA-1283 5ug Booster: Participants received a single booster dose of mRNA-1283 5 ug by intramuscular (IM) injection on day 1
- Part A: mRNA-1283 10ug Booster: Participants received a single booster dose of mRNA-1283 10 ug by intramuscular (IM) injection on day 1
- Part A: mRNA-1283.211 5ug Booster: Participants received a single booster dose of mRNA-1283.211 5 ug by intramuscular (IM) injection on day 1
- Part A: mRNA-1283.211 10ug Booster: Participants received a single booster dose of mRNA-1283.211 10 ug by intramuscular (IM) injection on day 1
- Part A: mRNA-1273 50ug Booster: Participants received a single booster dose of mRNA-1273 50 ug by intramuscular (IM) injection on day 1
- Part B: mRNA-1283.529 5ug Booster: Participants received a single booster dose of mRNA-1283.529 5 ug by intramuscular (IM) injection on day 1
- Part B: mRNA-1283.529 10ug Booster: Participants received a single booster dose of mRNA-1283.529 10 ug by intramuscular (IM) injection on day 1
Arm/Group | Part A: mRNA-1283 2.5ug Booster | Part A: mRNA-1283 5ug Booster | Part A: mRNA-1283 10ug Booster | Part A: mRNA-1283.211 5ug Booster | Part A: mRNA-1283.211 10ug Booster | Part A: mRNA-1273 50ug Booster | Part B: mRNA-1283.529 5ug Booster | Part B: mRNA-1283.529 10ug Booster
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/64 | 0/56 | 0/52 | 0/54 | 0/57 | 0/103 | 2/97
Serious Adverse Events (participants affected / at risk) | 2/57 | 1/64 | 2/56 | 3/52 | 3/54 | 2/57 | 2/103 | 6/97
Other Adverse Events (participants affected / at risk) | 15/57 | 13/64 | 16/56 | 18/52 | 12/54 | 16/57 | 24/103 | 24/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: mRNA-1283 2.5ug Booster (N=57) | Part A: mRNA-1283 5ug Booster (N=64) | Part A: mRNA-1283 10ug Booster (N=56) | Part A: mRNA-1283.211 5ug Booster (N=52) | Part A: mRNA-1283.211 10ug Booster (N=54) | Part A: mRNA-1273 50ug Booster (N=57) | Part B: mRNA-1283.529 5ug Booster (N=103) | Part B: mRNA-1283.529 10ug Booster (N=97)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: mRNA-1283 2.5ug Booster (N=57) | Part A: mRNA-1283 5ug Booster (N=64) | Part A: mRNA-1283 10ug Booster (N=56) | Part A: mRNA-1283.211 5ug Booster (N=52) | Part A: mRNA-1283.211 10ug Booster (N=54) | Part A: mRNA-1273 50ug Booster (N=57) | Part B: mRNA-1283.529 5ug Booster (N=103) | Part B: mRNA-1283.529 10ug Booster (N=97)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 8 (9) | 8 (11) | 5 (5) | 6 (9) | 6 (8) | 14 (15) | 17 (22)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT05137236/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT05137236/SAP_001.pdf